CLINICAL TRIAL: NCT06565858
Title: Can Cardiac Muscle Contraction Explain the Rarity of Tumors in the Heart?
Brief Title: Physical Activity and Sarcoma, Role and Impact on Outcome
Status: Not yet recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: L2-157
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-08

CONDITIONS: Sarcoma
Keywords: Sarcoma; Physical activity
MeSH Terms: conditions — Sarcoma; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to evaluate the role/impact of physical activity (PA) in sarcomas, in their distribution and potentially also on their prognosis, as already demonstrated for other neoplasms. Type, intensity, frequency, duration and circumstance of both occupational and leisure physical activity will be collected through validated questionnaires and self-reported measurement methods.

DETAILED DESCRIPTION:
The protective role of physical activity (PA) has been demonstrated in numerous diseases, especially cardiovascular and metabolic ones, but also in various neoplastic pathologies.

It has been estimated that approximately 25% of cancer cases globally are due to excess weight and a sedentary lifestyle. Regular moderate-intensity or greater physical activity is associated with a reduced risk of several types of cancer. Most studies have shown this association especially for breast, colon, and endometrial cancer.

The mechanisms through which PA may decrease cancer risk are numerous: physical activity might work through reducing the amount of adipose tissue, thereby lowering circulating levels of estrogens and other sex hormones, PA improves insulin resistance, reduces hyperinsulinaemia, might reduce inflammatory markers, thereby decreasing the exposure to these potentially carcinogenic hormones and peptides, reduces oxidative stress, reduces gastrointestinal transit time and improves immune system by increasing the phagocytic activity of macrophages and neutrophils, and increasing the proliferation of natural killer cells and lymphocytes. Other mechanisms under investigation pertain angiogenesis, DNA repair, and growth factors.

In addition to hormone-sensitive tumors and colon cancer, new evidence suggests that similar associations with PA might exist for other cancers for which less is known about the potential mechanisms underlying the physical activity association, suggesting that further mechanistic research is warranted.

Furthermore, in people who have already been diagnosed with cancer and are undergoing oncological therapy, regular exercise helps to counteract some typical and common side effects of anti-cancer therapies, thus improving treatment compliance and the overall quality of life. In particular, physical activity seems to reduce fatigue, arthralgia, nausea, improves cardiovascular and respiratory capacity, reduces the risk of osteoporosis, and anxiety.

Even more, several studies have shown that in patients already affected by cancer, physical activity could be associated with a better prognosis, reducing risk of recurrence and increasing survival. The most important and largest studies are mainly aimed at breast, colorectal, prostate and ovarian cancer [5-8].

Due to their rarity and extreme histological-molecular heterogeneity, little is known about sarcomas, particularly regarding potential risk factors and possible factors that may influence their clinical course.

Furthermore, starting from the evidence that cardiac tumors, both primary and secondary, are extremely rare, the possible mechanisms responsible for this favorable "refractoriness" of myocardial cells to neoplastic transformation and/or to the engraftment of other neoplastic cells will be studied.

The property of cardiomyocytes most likely related to this phenomenon is their contractility and continuous exposure to mechanical load that halt cardiomyocyte proliferation in the human heart. This project aims at improving knowledge about the molecular landscape and genetic aberrations involved in pathogenesis of cardiac tumors and assessing whether the mechanical forces generated by cardiomyocyte contraction in a beating heart inhibit the proliferation of cancer cells, thus protecting the heart from cancer.

Engineered heart tissue will be used to silence candidate mechanosensing genes. This should make the cell unresponsive to mechanical stimulation and thus allow it to proliferate even with increased afterload.

The expression levels of the mechanosensing genes eventually identified, will be tested in tumor tissue from sarcoma as located in the extremities of physically active individuals to assess whether they are downregulated, thus making the cells able to proliferate although located in actively contracting skeletal muscles.

Confirmation of the role of physical activity on cancer is awaited with interest. Understanding the mechanisms that link physical activity with cancer will be useful for several reasons. First, the identification of this mechanisms can give new clues to cancer biology, which might help in designing other cancer prevention and innovative treatment modalities. Second, if further data accumulate showing that increased physical activity can prevent some cancers or improve outcomes, this would constitute an excellent public health intervention to reduce the impact of cancer risks and costs.

ELIGIBILITY:
Inclusion Criteria:

* age >18;
* diagnose of sarcoma;
* Written informed consent must be signed and dated by the patient and the investigator.

Exclusion Criteria:

* Kaposi sarcoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective observational study recruiting patients diagnosed with sarcomas any site. Since sarcoma develop in bone, soft tissue and viscera, sarcoma appear suitable to investigate the role of physical activity on sarcoma in different locations.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence PA | 12 months
  The prevalence of physical activity (PA) in patients with sarcoma

CONTACTS AND LOCATIONS:
Overall Officials: Paola Queirolo, MD, Principal Investigator — Istituto Europeo di Oncologia
Locations (1):
- Istituto Europeo di Oncologia, Milan, Italy

REFERENCES:
- [Background] Meyerhardt JA, Heseltine D, Niedzwiecki D, Hollis D, Saltz LB, Mayer RJ, Thomas J, Nelson H, Whittom R, Hantel A, Schilsky RL, Fuchs CS. Impact of physical activity on cancer recurrence and survival in patients with stage III colon cancer: findings from CALGB 89803. J Clin Oncol. 2006 Aug 1;24(22):3535-41. doi: 10.1200/JCO.2006.06.0863. Epub 2006 Jul 5. PMID 16822843
- [Result] McTiernan A, Friedenreich CM, Katzmarzyk PT, Powell KE, Macko R, Buchner D, Pescatello LS, Bloodgood B, Tennant B, Vaux-Bjerke A, George SM, Troiano RP, Piercy KL; 2018 PHYSICAL ACTIVITY GUIDELINES ADVISORY COMMITTEE*. Physical Activity in Cancer Prevention and Survival: A Systematic Review. Med Sci Sports Exerc. 2019 Jun;51(6):1252-1261. doi: 10.1249/MSS.0000000000001937. PMID 31095082
- [Result] Matthews CE, Moore SC, Arem H, Cook MB, Trabert B, Hakansson N, Larsson SC, Wolk A, Gapstur SM, Lynch BM, Milne RL, Freedman ND, Huang WY, Berrington de Gonzalez A, Kitahara CM, Linet MS, Shiroma EJ, Sandin S, Patel AV, Lee IM. Amount and Intensity of Leisure-Time Physical Activity and Lower Cancer Risk. J Clin Oncol. 2020 Mar 1;38(7):686-697. doi: 10.1200/JCO.19.02407. Epub 2019 Dec 26. PMID 31877085
- [Result] Moore SC, Lee IM, Weiderpass E, Campbell PT, Sampson JN, Kitahara CM, Keadle SK, Arem H, Berrington de Gonzalez A, Hartge P, Adami HO, Blair CK, Borch KB, Boyd E, Check DP, Fournier A, Freedman ND, Gunter M, Johannson M, Khaw KT, Linet MS, Orsini N, Park Y, Riboli E, Robien K, Schairer C, Sesso H, Spriggs M, Van Dusen R, Wolk A, Matthews CE, Patel AV. Association of Leisure-Time Physical Activity With Risk of 26 Types of Cancer in 1.44 Million Adults. JAMA Intern Med. 2016 Jun 1;176(6):816-25. doi: 10.1001/jamainternmed.2016.1548. PMID 27183032
- [Result] McTiernan A. Mechanisms linking physical activity with cancer. Nat Rev Cancer. 2008 Mar;8(3):205-11. doi: 10.1038/nrc2325. PMID 18235448
- [Result] Ibrahim EM, Al-Homaidh A. Physical activity and survival after breast cancer diagnosis: meta-analysis of published studies. Med Oncol. 2011 Sep;28(3):753-65. doi: 10.1007/s12032-010-9536-x. Epub 2010 Apr 22. PMID 20411366
- [Result] Meyerhardt JA, Giovannucci EL, Ogino S, Kirkner GJ, Chan AT, Willett W, Fuchs CS. Physical activity and male colorectal cancer survival. Arch Intern Med. 2009 Dec 14;169(22):2102-8. doi: 10.1001/archinternmed.2009.412. PMID 20008694
- [Result] Meyerhardt JA, Giovannucci EL, Holmes MD, Chan AT, Chan JA, Colditz GA, Fuchs CS. Physical activity and survival after colorectal cancer diagnosis. J Clin Oncol. 2006 Aug 1;24(22):3527-34. doi: 10.1200/JCO.2006.06.0855. Epub 2006 Jul 5. PMID 16822844